CLINICAL TRIAL: NCT00441363
Title: A Randomized, Double-Blind, Parallel-Group Trial to Assess the Efficacy and Safety of Cycloset® Compared With Placebo When Added to Metformin in Patients With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of Cycloset® Compared With Placebo When Added to Metformin
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Failure to Recruit in a Timely manner
Sponsor: VeroScience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 165-AD-04-03-US-2
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-04

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Bromocriptine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bromocriptine Mesylate (Active Comparator): Bromocriptine mesylate 0.8 mg
  Interventions: Drug: Bromocriptine Mesylate
- Placebo (Placebo Comparator): Bromocriptine mesylate 0.8 mg matching placebo
  Interventions: Drug: Bromocriptine Mesylate

INTERVENTIONS:
Drug: Bromocriptine Mesylate — 0.8 mg tablet
  Other Names: Cycloset

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of Cycloset® and placebo when added to metformin monotherapy (at least 1000 mg/day for 3 months prior to screening) in persons with type 2 diabetes mellitus who are not adequately controlled on metformin therapy alone.

DETAILED DESCRIPTION:
In the previously conducted Phase III clinical trials, Cycloset® (up to a maximum dose of 4.8 mg/day), administered either as monotherapy or combined with sulfonylurea therapy, significantly reduced HbA1c, fasting and post-prandial glucose and fasting and post-prandial triglycerides in obese individuals with type 2 diabetes mellitus. Clinical studies that combined Cycloset® with metformin were not as part of the original Cycloset® clinical program because metformin was not commercially available in the United States at the time that the studies were initiated. The present study is designed to investigate the efficacy and safety of Cycloset® compared to placebo when added to metformin monotherapy in persons with type 2 diabetes mellitus who are not adequately controlled on metformin therapy alone.

A sufficient number of individuals will be screened to enroll up to 326 subjects;approximately 276 subjects are expected to complete treatment through study termination (Week 26). The study population will consist of individuals currently treated with metformin, for at least 3 months prior to the study start. Subjects who have ever received exogenous insulin therapy as part of an outpatient diabetes treatment regimen are to be excluded, as are those taking oral anti-diabetic agents other than metformin within 3 months of screening (e.g., sulfonylureas, thiazolidinediones,alpha-glucosidase inhibitors, or meglitinides). Subjects may be male or female(surgically sterile, postmenopausal, or using appropriate contraceptive methods if of childbearing potential), age 18 to 75 years, inclusive, and are to have a screening HbA1c value of ≥ 7.5% and <11.0% and a screening body mass index (BMI) in the range of 25 kg/m2 to 42 kg/m2, inclusive.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with type 2 diabetes mellitus, for at least six months prior to screening.
2. 18-75 years of age, inclusive.
3. Male or if female, is either:

   * postmenopausal or
   * of childbearing potential and has used appropriate contraceptive methods
4. Treated with a stable dose of metformin at least 3 months.
5. Has not been treated with a sulfonylurea, thiazolidinedione, meglitinide, alpha-glucosidase inhibitor, or combination oral anti-diabetic therapy within 3 months prior to screening.
6. Has not been on a regimen of lipid-lowering agents or if on such a regimen, it has been stable for a minimum of 6 weeks at screening.
7. HbA1c value between ≥ 7.5% and < 11%, at screening (Visit 1) and Visit 3.
8. Fasting plasma glucose measurement of ≤260 mg/dL at screening (Visit 1) and Visit 3.
9. Fasting C-peptide value equal to or greater than the normal accepted minimum value (e.g. < 0.9 NG/ml).
10. Stable body weight, i.e., not varying by > 10% for at least3 months prior to screening
11. Body mass index (BMI) at screening of 25 kg/m2 to 42 kg/m2,inclusive.
12. If treated for hypertension, the individual has been on stable therapy for 1 month prior to screening.

Exclusion Criteria:

1. Prior exogenous insulin therapy as part of an outpatient diabetes treatment regimen.
2. Type 1 diabetes mellitus
3. Clinically significant history of cardiac disease or presence of cardiac disease, including MI, clinically significant arrhythmia, unstable angina pectoris, moderate to severe congestive heart failure, CABG, or angioplasty; or expected to require CABG or angioplasty during the study.
4. Uncontrolled hypertension, defined as systolic blood pressure > 160 or diastolic blood pressure > 100 mmHg measured in sitting position at screening(Visit 1)

   Clinically significant history or presence of:
5. Hepatic disease (i.e. impaired liver function, including having AST or ALT greater than three times the upper limit of normal)
6. Renal disease (i.e. renal impairment with a serum creatinine ≥ 1.4 mg/dl)
7. Central nervous system disease, including epilepsy
8. CVA within the last 3 years.
9. Less than 5 years remission from clinically significant malignancy.
10. Major surgical operation within 3 months of screening.
11. Organ transplantation.
12. Evidence of acute or chronic illness including known or suspected HIV,HBV, or HCV infection.
13. Currently abuses drugs or alcohol, including binge drinking, or history of abuse that in the investigator's opinion would cause the individual to be noncompliant.
14. Regularly uses medications with addictive potential such as opiates,narcotics, tranquilizers, etc.
15. Used drugs for weight loss, e.g., Xenical® (orlistat), Meridia® (sibutramine),Acutrim® (phenylpropanolamine), or similar over-the-counter medications within 3 months of screening.
16. Known hypersensitivity to any components of the study drugs.
17. Received any experimental drug or used an experimental device within 3 months of screening or will do so during the study.
18. Has received unstable dose of fibric acid derivatives within 3 months of the screening.
19. Requires regular use of systemic corticosteroids by oral, intravenous (IV),or intramuscular (IM) route, or regular use of potent, inhaled intranasal steroids that are known to have a high rate of systemic absorption.
20. Prescription sympathomimetic drugs within 7 days of screening.
21. Started therapy with an erectile dysfunction drug within 2 weeks prior to screening. The subject may not begin treatment with an erectile dysfunction drug during the study period; subjects previously taking erectile dysfunction drugs should do so only under medical supervision.
22. Donated blood within 60 days of screening. Donation of blood also is prohibited during the study and for 30 days after completion of the study.
23. Occupation that requires a rotation of shift work or working over night shifts.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2005-02; Primary Completion 2006-02 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Scranton, MD, Study Director — VeroScience

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was originally designed to enroll 326 subjects in order to randomize 225 subjects. Due to a strategic business decision of the former sponsor (PLIVA), enrollment into the study was prematurely terminated.
Groups:
- Cycloset: 0.8 mg tablet
- Placebo: matching placebo
Period: Overall Study
Arm/Group | Cycloset | Placebo
Started | 32 | 34
Completed | 15 (no subject withdrew early since the trial was terminated) | 19
Not Completed | 17 | 15
Not completed — Adverse Event | 4 | 2
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Physician Decision | 6 | 7
Not completed — Lost to Follow-up | 2 | 2
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cycloset | Placebo | Total
Number analyzed (Participants) | 32 | 34 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (10.5) | 53 (9.3) | 53 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 17 | 20 | 37
Region of Enrollment [Number; unit: participants]
  United States | 32 | 34 | 66

OUTCOME MEASURES:

1. Primary Outcome: Change in Baseline to End of Study in HbA1c
Description: Too few subjects were enrolled to assess outcome to pre-specified statistical power.
Time Frame: up to 24 weeks
Measure: Mean (Standard Deviation); unit: % HbA1c
Arm/Group | Cycloset | Placebo
Number analyzed (Participants) | 32 | 34
% HbA1c | -0.4 (.95) | -.5 (0.87)

2. Secondary Outcome: Fasting Plasma Glucose and Lipids
Time Frame: up to 24 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Number of Serious Adverse Events Experienced by the Subjects
Time Frame: up to 24 weeks
Population: Report of Serious adverse events that occurred in the trial.
Measure: Number; unit: serious adverse events
Arm/Group | Cycloset | Placebo
Number analyzed (Participants) | 32 | 34
serious adverse events | 1 | 0

ADVERSE EVENTS:
Arm/Group | Cycloset | Placebo
Serious Adverse Events (participants affected / at risk) | 1/32 | 0/34
Other Adverse Events (participants affected / at risk) | 20/32 | 14/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cycloset (N=32) | Placebo (N=34)
unstable angina (Cardiac disorders) | 1 (1) | 0 (0) — The only SAE in the study was reported in a subject from the Cycloset™ treatment group who experienced unstable angina and dyspnea. Both events were deemed by the site investigator as unlikely related to study drug and resolved.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cycloset (N=32) | Placebo (N=34)
nausea (Gastrointestinal disorders) | 6 | 3
vomiting (Gastrointestinal disorders) | 3 | 2
Urinary Tract Infection (Infections and infestations) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 2
Vision blurred (Eye disorders) | 2 | 0
Fatigue (General disorders) | 2 | 0
Sinusitis (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes